CLINICAL TRIAL: NCT04303572
Title: Phase III Multi-Center, Randomized, Controlled Inhibitor Eradication Trial, Comparing Eloctate Immune Tolerance Induction (ITI) Plus Emicizumab vs. Eloctate ITI Alone to Eradicate Inhibitor Formation in Severe Hemophilia A
Brief Title: The Hemophilia Inhibitor Eradication Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The INHIBIT Trials IDSMB, in a letter dated 05-18-22, recommended, given the slow enrollment, that the INHIBIT Trials be discontinued due to futility.
Sponsor: Margaret Ragni (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Margaret Ragni, Professor of Medicine and Clinical and Translational Research, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO19070080; H30MC24050 (Other Grant/Funding Number: (HRSA) Health Resources and Services Administration)
Record Dates: First submitted 2019-10-31; First posted 2020-03-11 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Hemophilia A With Inhibitor
Keywords: hemophilia; inhibitor formation; Eloctate; Emicizumab
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein; emicizumab

STUDY DESIGN:
Intervention Model Description: This is a phase III open-label, randomized controlled trial comparing immune tolerance induction with one drug, with or without a second drug in the eradication of hemophilia inhibitors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eloctate ITI plus Emicizumab (Experimental): Arm A: Eloctate 100 IU/kg every other day by intravenous infusion plus Emicizumab 1.5 mg/kg subcutaneously (following 3 mg/kg/wk x 4 induction) in children and adults with severe hemophilia A and anti-FVIII inhibitor, continued up to 48 weeks.
  Interventions: Drug: Eloctate ITI; Drug: Emicizumab
- Eloctate ITI (Active Comparator): Arm B: Eloctate 100 IU/kg every other day by intravenous infusion in children and adults with severe hemophilia A and anti-FVIII inhibitor, continued up to 48 weeks.
  Interventions: Drug: Eloctate ITI

INTERVENTIONS:
Drug: Eloctate ITI — This is a factor VIII-Fc infusion protein.
  Other Names: rFVIIIFc
Drug: Emicizumab — This is a bispecific monoclonal antibody FVIII mimic.
  Other Names: Hemlibra
  Arms: Eloctate ITI plus Emicizumab

SUMMARY:
This is a multi-center randomized phase III clinical trial, the Inhibitor Eradication Trial, in which Eloctate ITI plus Emicizumab will be compared with Eloctate ITI alone to eradicate inhibitors in severe hemophilia A.

DETAILED DESCRIPTION:
This is a multi-center randomized phase III clinical trial, the Inhibitor Eradication Trial, in which Eloctate ITI plus Emicizumab will be compared with Eloctate ITI alone to eradicate inhibitors in patients with severe hemophilia A This adaptive design is necessary as randomized trials in rare diseases are often not possible. The INHIBIT Clinical Trials Platform includes two linked trials, the Inhibitor Prevention Trial (Prevention Trial) and the Inhibitor Eradication Trial (Eradication Trial) that will be conducted at up to 41 U.S. hemophilia treatment centers (HTCs) affiliated with universities. The Inhibitor Eradication Trial is a 48-week randomized phase III trial, in which 90 previously treated patients (PTPs) with severe hemophilia A and high-responding inhibitors (anti-VIII > 0.6 B.U.), will be enrolled. Subjects will include individuals with severe hemophilia A who develop inhibitors during the linked Inhibitor Prevention Trial and adults or children at the same HTCs refractory to or never undergoing immune tolerance induction (ITI). Once enrolled, subjects who meet all the inclusion and none of the exclusion criteria, will be randomized to weekly Eloctate ITI plus weekly Emicizumab vs. weekly Eloctate ITI alone to eradicate inhibitor formation, defined as anti-FVIII<0.6 B.U. Blood draws will be minimized to 6 timepoints, pre, 4, 12, 24, 36, and 48 weeks, and validated for small volumes, 3.8 cc (¾ tsp) each. The Inhibitor Eradication Trial is considered greater than minimal risk as study drug is given before the first bleed and special inhibitor studies are obtained. (NB: The Inhibitor Eradication Trial (PRO19070080) is linked to the Inhibitor Prevention Trial (PRO19040140), as part of the INHIBIT Clinical Trials Platform, and both trials will be conducted efficiently in the same hemophilia treatment centers (HTCs), with the same MDs, coordinators, visit frequency, blood sampling, and assays.

ELIGIBILITY:
Inclusion Criteria:

1. Male adults or children > 4 months of age.
2. Severe hemophilia A (FVIII < 0.01 U/ml).
3. Current or past high-responding inhibitor, anti-FVIII >= 5.0 B.U., ITI-refractory or ITI-naive.

Exclusion Criteria:

1. Acquired hemophilia or any bleeding disorder other than hemophilia A.
2. Current use of Emicizumab, or if used, > 8 weeks since last treatment.
3. Use of an experimental drug(s).
4. Surgery anticipated in the next 48 weeks.
5. Life expectancy less than 5 years.
6. Patient/parent/caretaker unable or unwilling to keep a personal diary of bleeding frequency and study drug treatment, make monthly visits and blood draws at weeks 4, 8, 12, 24, 36, and 48.
7. Other illness, condition, or reason in the opinion of the investigator that would make the patient unsuitable for the trial.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret V Ragni, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Hemophilia Center of Western PA, Pittsburgh, Pennsylvania
  - University of Pittsburgh and Hemophilia Center Western PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
A biologic specimen and data repository for this trial will be available at the Graduate School of Public Health (GSPH) Data Center repository for investigators who make formal application request and is formally approved by the Coordinating Center (Pitt) and Data Center (GSPH).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one year of trial completion.
Access Criteria: Access will be determined by the Study Team.

REFERENCES:
- [Background] Ragni MV, George LA; Members of Working Group 1, the NHLBI State of the Science Workshop on factor VIII inhibitors: Generating a national blueprint for future research. The national blueprint for future factor VIII inhibitor clinical trials: NHLBI State of the Science (SOS) Workshop on factor VIII inhibitors. Haemophilia. 2019 Jul;25(4):581-589. doi: 10.1111/hae.13717. PMID 31329364
- [Background] Ebbert PT, Xavier F, Malec LM, Seaman CD, Ragni MV. Observational study of recombinant factor VIII-Fc, rFVIIIFc, in hemophilia A. Thromb Res. 2020 Nov;195:51-54. doi: 10.1016/j.thromres.2020.07.004. Epub 2020 Jul 5. PMID 32653601
- [Background] Bertolet M, Brooks MM, Ragni MV. The design of a Bayesian platform trial to prevent and eradicate inhibitors in patients with hemophilia. Blood Adv. 2020 Nov 10;4(21):5433-5441. doi: 10.1182/bloodadvances.2020002789. PMID 33156923

RESULTS

PARTICIPANT FLOW:
Groups:
- Eloctate ITI: Eloctate 100 IU/kg every other day by intravenous infusion in children and adults with severe hemophilia A and anti-FVIII inhibitor, continued up to 48 weeks.
  Eloctate ITI: This is a factor VIII-Fc infusion protein.
Period: Overall Study
Arm/Group | Eloctate ITI
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study closed due to poor enrollment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eloctate ITI
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 1 [1 to 1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
Number and Type of Bleeds in the last year [Number; unit: Bleeds] | 0
Prior Circumcision [Count of Participants; unit: Participants] | 1
Anti-FVIII level > 0.6 BU [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Inhibitor Eradication
Description: The proportion eradicating anti-FVIII inhibitors
Time Frame: 48 weeks
Population: Only patient was enrolled on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Eloctate ITI
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Number of Bleeding Events
Description: The number of bleeding events: hematoma, joint, central nervous system, other bleeds.
Time Frame: 48 weeks
Population: Only patient was enrolled on study.
Measure: Number; unit: number of bleeding events
Arm/Group | Eloctate ITI
Number analyzed (Participants) | 1
number of bleeding events | 0

3. Secondary Outcome: FVIII Trough Level
Description: The FVIII trough activity by chromogenic assay.
Time Frame: 48 weeks
Population: specimen collected, discarded with out analysis due to study being close dearly due to low enrollment
Arm/Group | Eloctate ITI
Number analyzed (Participants) | 0

4. Secondary Outcome: Human Leukocyte Antigen (HLA) Haplotype
Description: The number of HLA haplotype variants.
Time Frame: 48 weeks
Population: specimen collected, discarded with out analysis due to study being close dearly due to low enrollment
Arm/Group | Eloctate ITI
Number analyzed (Participants) | 0

5. Secondary Outcome: FVIII Mutation
Description: The number of FVIII mutation variants.
Time Frame: 48 weeks
Population: specimen collected, discarded with out analysis due to study being close dearly due to low enrollment
Arm/Group | Eloctate ITI
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: Adverse events were self-reported.
Arm/Group | Eloctate ITI
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT04303572/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT04303572/ICF_002.pdf